CLINICAL TRIAL: NCT04888767
Title: Assessment of the Safety and Feasibility of a High-intensity Interval Training Program in Adult CF Patients: a Randomized Bicentric Pilot Study
Brief Title: Safety and Feasibility of High-intensity Interval Training Program in CF Patients
Acronym: ITHI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ildys (Other)
Collaborators: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILDYS-ISC2-2020-002; ID-RCB (Other: 2021-A00512-39)
Record Dates: First submitted 2021-05-06; First posted 2021-05-17 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Respiratory rehabilitation program; Physical activity; High intensity interval training; Quality of life
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity

STUDY DESIGN:
Intervention Model Description: * Bicentric; prospective; opened ; randomized; controlled study
  * Distribution of patients in groups according to a ratio (1:1)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients benefiting from the usual re-training sessions
- ITHI Group (Experimental): Patients benefiting from ITHI re-training sessions
  Interventions: Other: Interval Training Hight Intensity Program

INTERVENTIONS:
Other: Interval Training Hight Intensity Program — * Rehabilitation stay in hospitalization with 18 days of training sessions
  * Training on an ergometer
  * Sessions supervised by an Adapted Physical Activities (APA) teacher or a physiotherapist
    * Control group: 5 times / week; continuous work 20 to 30 min; around the 1st aerobic ventilation threshold
    * Intervention group: 2 times / week: maintenance sessions + 3 times / week: IHTI sessions - alternating 30s work / 30s rest repeated 6 times; at 60% of the maximum heart rate at the 1st session then increase as fast and large as possible
  Arms: ITHI Group

SUMMARY:
This study compare an usual training program (in continuous endurance) with an ITHI program over a period of 3 weeks, in France. The aim is to evaluate the safety and feasibility of this type of program in CF adults, and also more specifically, in subgroups:

patients divided according to the severity of their FEV1 ; patients treated with modulating CFTR canal therapy ; diabetic patients on insulin ; undernourished patients.

DETAILED DESCRIPTION:
Objectives Studies have shown good tolerance of High Intensity Interval Training (ITHI) in healthy people or in COPD with similar results obtained with continuous training regimen, but with less shortness of breath and muscle fatigue, greater pleasure and a positive impact on glycemia. Research in CF is still scarce.

We propose to compare our usual training program (in continuous endurance) with an ITHI program over a period of 3 weeks, corresponding to the length of the rehabilitation stay in France. Our aim is to evaluate the safety and feasibility of this type of program in CF adults, and also more specifically, in subgroups:

* patients divided according to the severity of their FEV1
* patients treated with modulating CFTR canal therapy
* diabetic patients on insulin
* undernourished patients (BMI ≤ 18.5)

Methodology

* Bicentric (Roscoff-Giens); prospective; opened; randomized; controlled
* Rehabilitation stay in hospitalization with 18 days of training, on an ergometer, supervised by an APA teacher or a physiotherapist

  * Control group: 5 times / week; continuous work 20 to 30 min; around the 1st aerobic ventilation threshold
  * Intervention group: 2 times / week: maintenance sessions + 3 times / week: IHTI sessions - alternating 30s work / 30s rest repeated 6 times; at 60% of the maximum heart rate at the 1st session then increase as fast and large as possible
* Distribution of the 100 patients included in a 1: 1 ratio
* Examinations / Questionnaires in current practice: medical consultation; quality of life (CFQ-R); anxiety-depression (HAD); "Starfish" (Feelings linked to physical activity) ; blood sugar (Freestyle); impedance measurement; respiratory capacity measurement ; Voluntary Driving Force; walk test (TM6); dyspnea scale (Borg)
* Study-specific measures: MDP (Multidimensional Profile of Dyspnea) and PACES (Physical Activity Enjoyment Scale) scales

Expected results

Through this pilot study we are expecting to answer several questions:

* are the safety and tolerance of an ITHI program at least equal if not better than that of a "classic" training?
* what about the most severe patients?
* could patients on modulator have ITHI training (treatment likely to increase creatine kinase - muscle enzyme -)?
* are diabetic patients more at risk of hypoglycaemia during an ITHI compared to traditional training?
* could undernourished patients participate in ITHI regimen?

Perspective If ITHI appears to be safe and well tolerated, it could be integrated into "classic" rehabilitation programs and represent an interesting alternative, depending on the profile of each patient. The effectiveness of the ITHI program will also be discussed by evaluating several parameters, including 6mn walking distance test (6MWD). The emerging trends would allow some recommendations and more in-depth studies.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged over 18 years of age on the date of informed consent
* diagnosed CF patients
* not transplanted and not on the transplant waiting list
* able to participate in the proposed training programs (especially without cardiac contraindication)
* able to understand and respect the protocol and its requirement
* who signed the consent prior to any other procedure protocol

Exclusion Criteria:

* major patients under guardianship / curatorship / legal protection
* pregnant patients
* dialysis patients
* patients with a severe exacerbation at the time of inclusion
* patients for whom a new modulating treatment (eg.: Kaftrio®, Kalydeco®, Symkevi®, etc.) has been implemented in the 4 weeks preceding inclusion
* patients with pulmonary arterial hypertension (≥ 25 mmHg)
* patients unable to complete the entire program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Feasability evaluation | Continuous measurement over the entire stay (Day 1 to Day 18)
  Proportion of sessions carried out according to the planned program (and, in parallel, number and reasons for stopping sessions or the program)
Tolerance evaluation | Change from baseline (Day 2) at 3 weeks (Day 18)
  Scores on the Borg scale (physical activity dyspnea and muscle fatigue) : 0 to 10 - Higher score = worse outcome

SECONDARY OUTCOMES:
Cystic Fibrosis Questionnaire Revised (CFQR) | Change from baseline (Day 2) at 3 weeks (Day 18)
  Scores on CFQR (assessment of quality of life) : 0 to 100 - Higher score = better outcome
Hospital Anxiety and Depression scale (HAD) | Change from baseline (Day 2) at 3 weeks (Day 18)
  Scores on HAD : 2 scores (1 for anxiety and 1 for depression) - 0 to 21 - Higher score = worse outcome
Starfish | Change from baseline (Day 2) at 3 weeks (Day 18)
  Scores on the "starfish": assesment of the feelings about physical activity with an educational diagram - 12 "branches" = 12 sub-scores - 0 to 12 - Higher score = better outcome
Anthropometry | Change from baseline (Day 1) at 3 weeks (Day 18)
  Weight (Kg) and height (cm) will be combined to report BMI in kg/m2
Continuous blood sugar levels | Continuous measurement over the entire stay (Day 1 to Day 18)
  Evaluation of the glucose levels (average, minimum, maximum)
Ponctual blood sugar levels | Measurement at each sessions from Day 2 to Day 18
  Blood glucose assessment during re-training sessions (at the start; during; at the end; after recovery)
Impedance | Change from baseline (Day 2) at 3 weeks (Day 18)
  Bioelectrical impedance analysis of body composition
Spirometry | Change from baseline (Day 2) at 3 weeks (Day 18)
  Respiratory capacity assessment : forced expiratory volume in 1 second (FEV1)
Maximal Voluntary force : Strength | Change from baseline (Day 2) at 3 weeks (Day 18)
  Best measurement, in Newton, of thigh quadriceps strength after 6 evaluations (3 with the left thigh and 3 with the right thigh)
Maximal Voluntary force : endurance | Change from baseline (Day 2) at 3 weeks (Day 18)
  Best measurement, in second, of thigh quadriceps strength after 2 evaluations (13 with the left thigh and 1 with the right thigh)
6MWT | Change from baseline (Day 12) at 3 weeks (Day 18)
  Measurement of the distance traveled during the six minutes walk test (6MWT) and of several related parameters (dyspnea, oxygen saturation, heart rate - at the start, at the finish, after rest)
Multidimensional dyspnea profile scale (MDP) | Change from baseline (Day 2) at 3 weeks (Day 18)
  Scores on the MDP : assessment of discomfort (0 to 10), sensory component (0 to 50) and affective component (0 to 50) of breathlessness -> 3 sub-scores - Higher score = worse outcome
Physical Activity Enjoyment Scale (PACES) | Measurement at the end of the stay (Day 18)
  Score on the PACES : assessment of global satisfaction felt during re-training sessions - 10 to 70 - Higher score = better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Ramel, MD, Principal Investigator — Fondation Ildys
Locations (2):
- France (2):
  - CF Center - Fondation Ildys Site de Perharidy, Roscoff, Finistère
  - CF Center of Giens - Hospices Civils de Lyon Hôpital Renée Sabran, Giens, Hyères

IPD SHARING:
Plan to Share IPD: No